CLINICAL TRIAL: NCT03508193
Title: Reverse-Engineering of Exclusive Enteral Nutrition (RE-EEN) in Crohn's Disease
Brief Title: Reverse Engineering of Exclusive Enteral Nutrition
Acronym: RE-EEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dale Lee (Other)
Responsible Party: Sponsor-Investigator, Dale Lee, Associate Professor of Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000619
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Crohn Disease
Keywords: Exclusive Enteral Nutrition; Nutrition; Diet; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Whole-foods based smoothie as nutritional therapy
  Interventions: Other: Nutritional therapy

INTERVENTIONS:
Other: Nutritional therapy — Whole-foods based smoothie designed to emulate formulas used in EEN

SUMMARY:
Primary: Nutritional therapy in the form of a whole-food based smoothie can be used to induce remission of active Crohn's disease.

Secondary: Consuming a whole foods based smoothie will result in measurable changes to the microbiome of individuals with Crohn's disease and healthy controls.

The specific aims of this proposal are:

1. To develop a whole-food based smoothie, based on principles of the specific carbohydrate diet, that is comparable in macronutrients and micronutrients to formulas used for exclusive enteral nutritional (EEN) therapy in Crohn's disease.
2. To evaluate the ability of a whole-food based smoothie to induce remission of active Crohn's disease.
3. To evaluate changes to the intestinal microbiome in healthy individuals consuming a whole-food based smoothie diet.

DETAILED DESCRIPTION:
This will be an open label, pilot study over 4 weeks in children with newly diagnosed Crohn's disease treated with a smoothie designed to emulate formulas used for exclusive enteral nutritional therapy. In place of formula, whole-foods based smoothie recipes and the food to create the smoothies will be given to each participant/family. The smoothies will be based upon the concept of reverse-engineering of exclusive enteral nutrition (RE-EEN). The smoothie recipes will involve whole foods that can be blenderized to liquid consistency. Similar to the formulas used for EEN, the smoothies will provide calories, protein, fat, and carbohydrates in a distribution to support growth and development.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 -21 years old
2. Diagnosis of Crohn's disease within 4 weeks of study entry
3. Active Crohn's disease, as defined by Pediatric Crohn's Disease Activity Index (PCDAI) ≥10.
4. Participant capable of giving informed consent, or if a minor the parent/guardian is capable of giving informed consent

Exclusion Criteria:

1. History of surgery for Crohn's disease
2. Perianal disease as part of Crohn's disease phenotype
3. Prior treatment with EEN or the specific carbohydrate for Crohn's disease
4. Prior treatment with any immunosuppressive medication (corticosteroids, anti-TNF-alpha agent, azathioprine, methotrexate, etc.)
5. Prior treatment with antibiotics for Crohn's disease
6. Known allergies to any of the food components in the smoothie
7. Admission to hospital due to severity of Crohn's disease and associated symptoms
8. Unwillingness to provide informed consent

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Fecal calprotectin <250 micrograms/gram | 4 weeks
  surrogate marker of intestinal inflammation

SECONDARY OUTCOMES:
Quality of life as measured by IMPACT III Questionnaire | 4 weeks
  validated quality of life measure for pediatric inflammatory bowel disease

CONTACTS AND LOCATIONS:
Overall Officials: Dale Y Lee, MD, Principal Investigator — Seattle Children's Hospital and The University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Not Discussed

REFERENCES:
- [Background] Johnson T, Macdonald S, Hill SM, Thomas A, Murphy MS. Treatment of active Crohn's disease in children using partial enteral nutrition with liquid formula: a randomised controlled trial. Gut. 2006 Mar;55(3):356-61. doi: 10.1136/gut.2004.062554. Epub 2005 Sep 14. PMID 16162683
- [Background] Lee D, Baldassano RN, Otley AR, Albenberg L, Griffiths AM, Compher C, Chen EZ, Li H, Gilroy E, Nessel L, Grant A, Chehoud C, Bushman FD, Wu GD, Lewis JD. Comparative Effectiveness of Nutritional and Biological Therapy in North American Children with Active Crohn's Disease. Inflamm Bowel Dis. 2015 Aug;21(8):1786-93. doi: 10.1097/MIB.0000000000000426. PMID 25970545
- [Derived] Lee D, Braly K, Nuding M, Braly I, Hopp C, Twible H, Pope C, Hayden HS, Hoffman L, Zheng H, Wahbeh G, Suskind DL. Reverse-engineered exclusive enteral nutrition in pediatric Crohn's disease: A pilot trial. J Pediatr Gastroenterol Nutr. 2024 May;78(5):1135-1142. doi: 10.1002/jpn3.12196. Epub 2024 Apr 1. PMID 38558411